CLINICAL TRIAL: NCT00910156
Title: Indirect Versus Direct Laryngoscopy for Routine Nasotracheal Intubation: a Pilot Study
Brief Title: Indirect Laryngoscopy for Nasal Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: General Hospital Linz (Other)
Other Study IDs: P01
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Intubation, Intratracheal

ARMS (3):
- Airtraq (Active Comparator)
  Interventions: Device: Airtraq laryngoscope
- Glidescope (Active Comparator)
  Interventions: Device: Glidescope laryngoscope
- Macintosh (Active Comparator)
  Interventions: Device: Macintosh laryngoscope

INTERVENTIONS:
Device: Airtraq laryngoscope — Airtraq intubation
  Arms: Airtraq
Device: Glidescope laryngoscope — glidescope intubation
  Arms: Glidescope
Device: Macintosh laryngoscope — Macintosh intubation
  Arms: Macintosh

SUMMARY:
Comparison of ease and convenience of nasotracheal intubation with the use of the two indirect laryngoscopes, Airtraq or Glidescope, versus the traditionally used Macintosh laryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* nasotracheal intubation

Exclusion Criteria:

* anticipated difficult airway
* risk factors for gastric aspiration
* history of bleeding
* relevant allergy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Intubation Difficulty Scale (IDS)

SECONDARY OUTCOMES:
Posture of the intubator

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital Linz, Linz, Austria